CLINICAL TRIAL: NCT01233401
Title: Tdap Vaccination for Infant Caregivers in the Pediatric Office
Brief Title: Tdap Vaccination for Infant Caregivers
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Saint Raphael Healthcare System (Other)
Responsible Party: Deepa Camenga, MD, Yale University
Other Study IDs: 1005006837
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Pertussis; Vaccination
Keywords: Pertussis, Vaccination, Adult
MeSH Terms: conditions — Whooping Cough | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mothers
  Interventions: Other: Survey
- Other Infant Caregivers: Includes fathers, grandparents, and other adults who are infant caregivers
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Mothers and Other infant caregivers are surveyed at the end of the 2 week newborn well child visit about whether they chose to receive the Tdap vaccine at the pediatrician's office.

SUMMARY:
This study evaluates whether offering Tetanus, diphteria and acellular pertussis (Tdap) vaccine to caregivers of newborn infants during pediatric well child visits increase the caregivers' vaccination rates.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* English or Spanish speaking

Exclusion Criteria:

* Do not speak English or Spanish

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18-64 year old men and women who are mothers or other infant caregivers of 2 week old infants
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maternal Tdap Vaccination Rate | At 2 week well child visit

SECONDARY OUTCOMES:
Other Infant Caregiver Tdap Vaccination Rate | At 2 week well child visit

CONTACTS AND LOCATIONS:
Overall Officials: Deepa R Camenga, MD, Principal Investigator — Yale University; Marjorie Rosenthal, MD MPH, Principal Investigator — Yale University
Locations (1):
- Hospital of St. Raphael, New Haven, Connecticut, United States